CLINICAL TRIAL: NCT01046357
Title: A Randomized, Blind, Placebo-controlled, Single-centre Phase I Study in Healthy Volunteers to Assess the Safety, Tolerability and Pharmacokinetics of AZD7687 After Single Ascending Oral Doses
Brief Title: A Study in Healthy Volunteers to Assess the Tolerability and Blood Levels of a Single Dose of AZD7687
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D2710C00001
Record Dates: First submitted 2009-12-03; First posted 2010-01-12 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: First in human; Safety
MeSH Terms: interventions — AZD7687

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): AZD7687 oral suspension
  Interventions: Drug: AZD7687
- Placebo (Experimental): placebo oral suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7687 — Single oral dose
  Arms: Active
Drug: Placebo — Single oral dose
  Arms: Placebo

SUMMARY:
This is a Phase I, first time in human, randomised, blinded, placebo-controlled, single ascending dose study in healthy male volunteers conducted at a single centre. The effect of food on the pharmacokinetics of AZD7687 will also be studied.

The study will consist of two parts, a dose escalation part and a food interaction part. The two parts will be run in parallel. In total, 64 healthy volunteers divided in 8 different panels (8 volunteers per cohort) will be exposed to single doses during the dose escalation. Each subject will receive dose only once, except for the volunteers included in the dose steps repeated for food interaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI between 19-30

Exclusion Criteria:

* No blood donation prior 30 days
* No other clinical study prior 3 months

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examination, telemetry, digital electrocardiograms (dECGs), safety 12-lead paper electrocardiograms (pECG), and clinical laboratory assessments)

SECONDARY OUTCOMES:
Plasma concentrations of AZD7687 and plasma pharmacokinetic parameters.
Exploratory pharmacogenetic blood sampling.
Pharmacodynamic biomarker sampling; blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States